CLINICAL TRIAL: NCT01461330
Title: Lifestyle Changes in Patients With Type 2 DM and Hypertension: DASH Diet and Exercise Effects
Brief Title: Lifestyle Changes in Patients With Type 2 Diabetes Mellitus and Hypertension
Status: Terminated | Phase: Not Applicable | Type: Interventional
Sponsor: Hospital de Clinicas de Porto Alegre (Other)
Responsible Party: Principal Investigator, Mirela Jobim de Azevedo, Dr., MD, Associated Professor of Medicine, Hospital de Clinicas de Porto Alegre
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: HCPA 10-0411
Record Dates: First submitted 2011-08-03; First posted 2011-10-28 (Estimated); Last update posted 2017-01-26 (Estimated); Status verified 2017-01

CONDITIONS: Blood Pressure
Keywords: diabetes; exercise; DASH diet; ABPM
MeSH Terms: conditions — Diabetes Mellitus; Motor Activity | interventions — Dietary Approaches To Stop Hypertension; Exercise

STUDY DESIGN:
Intervention Model Description: intervention: DASH diet plus exercise DASH diet adapted to the usual diet of Brazilian type 2 diabetic patients = prescription of a normocaloric diet including fruits, vegetables, grain products, low fat dairy foods, legumes, without sugar, and with limited fat Exercises: the recommended physical activity will consist of using a pedometer during the experimental period.
  active comparator = ADA diet = Adoption of ADA diet.
Oversight: Data Monitoring Committee: No

ARMS (2):
- DASH diet (Experimental): DASH DIET + EXERCISE
  Interventions: Other: DASH diet plus exercise
- ADA DIET (Active Comparator): DIET ACCORDING AMERICAN DIABETES ASSOCIATION DIETARY RECOMMENDATIONS FOR DIABETES
  Interventions: Other: ADA diet

INTERVENTIONS:
Other: DASH diet plus exercise — DASH diet adapted to the usual diet of Brazilian type 2 diabetic patients = prescription of a normocaloric diet including fruits, vegetables, grain products, low fat dairy foods, legumes, without sugar, and with limited fat
  Exercises: the recommended physical activity will consist of using a pedometer during the experimental period.
  Other Names: LYFESTYLE INTERVENTION
  Arms: DASH diet
Other: ADA diet — Adoption of ADA diet.
  Other Names: Active comparator: ADA DIET
  Arms: ADA DIET

SUMMARY:
Data obtained in hypertensive patients without diabetes suggest that increased association of non-pharmacological treatment in patients with diabetes and hypertension may be associated with an improvement in blood pressure control. Despite the beneficial results found, is not yet known the magnitude of the effect of a DASH diet associated with the stimulus of physical activity on BP in patients with type 2 diabetes. The beneficial effects on blood pressure of an additional non-pharmacological intervention to drug therapy may have an even greater impact in patients with treatment-resistant hypertension The aim of this study is to evaluate the effect of changes in lifestyle on blood pressure in patients with type 2 diabetes and hypertension resistant to treatment.

DETAILED DESCRIPTION:
The aim of this study is to evaluate the effect of changes in lifestyle on blood pressure in patients with type 2 diabetes and hypertension. Secondary objectives are: Assess whether the prescription of a DASH-type diet and encouragement for physical activity through use of pedometers, can improve blood pressure control in patients with type 2 diabetes and hypertension resistant to treatment.

Forty type 2 diabetic with resistant hypertension outpatients were included in a randomized clinical trial: treatment 1- DASH diet + encouragement for physical activity through use of pedometer; treatment 2- ADA diet + usual exercises. The duration of each treatment are four weeks. The patients included should have performed Ambulatory Blood Pressure Monitoring (ABPM) to exclude white-coat effect, ie when there are abnormal in the measurement of office blood pressure (equal to or above 140/90 mm Hg) and normal blood pressure by ABPM during the awake period (equal to or below 135/85 mm Hg). Twenty-four hour records with concurrent 24h urinary collections (protein intake estimative), clinical and laboratory evaluation were performed at baseline and after 4 weeks. Serum fatty acids were measured in total lipids by gas chromatography.

ELIGIBILITY:
Patients

Inclusion Criteria:

* type 2 diabetes
* Blood pressure ≥140/90 mm Hg
* ABMP ≥ 135/85 mm Hg

Exclusion Criteria:

* digestive disease with malabsorption
* diabetic neuropathy with gastroparesis
* BMI ≥ 40 kg/m²

Ages: 30 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2011-02 (Actual); Primary Completion 2013-10 (Actual); Study Completion 2013-11 (Actual)

PRIMARY OUTCOMES:
Change from Baseline in Blood Pressure at 4 weeks | 4 weeks
  Ambulatory Blood Pressure Monitoring (ABPM) at baseline and after 4 weeks

SECONDARY OUTCOMES:
Change from Baseline in glucose control at 4 weeks | 4 weeks
  A1 C test at baseline and after 4 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Tatiana P de Paula, RD, Study Chair — Hospital de Clínicas de Porto Alegre; Luciana Verzoça, MD, Study Chair — Hospital de Clínicas de Porto Alegre
Locations (1):
- Hospital de Clínicas de Porto Alegre, Porto Alegre, Rio Grande do Sul, Brazil